CLINICAL TRIAL: NCT03269370
Title: Randomized Controlled Trial of a Family-focused CBT Skills App and Standard Self Help Options for Childhood Anxiety and Related Conditions
Brief Title: Family-Focused CBT Skills App and Standard Self Help Options for Childhood Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas City Center for Anxiety Treatment, P.A. (Industry)
Collaborators: Virtually Better, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2R44MH098470-03 (NIH)
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Anxiety Disorders; Childhood Mental Disorder; Anxiety
Keywords: CBT; Self-Help; Family
MeSH Terms: conditions — Anxiety Disorders; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: RCT with 4 arms, one being a waitlist arm that allows for re-randomization into one of the 3 "active" study arms.
Masking Description: There is no masking in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1: Anchors Away (Experimental): Family will receive access to the basic Anchors Away mobile app to test over 6 weeks.
  Interventions: Behavioral: Anchors Away
- 2: Parent Enhanced Anchors Away (Experimental): Family will receive access to the Parent Enhanced Anchors Away mobile app to test over 6 weeks.
  Interventions: Behavioral: Parent Enhanced Anchors Away
- 3: Self-Help E-Book (Active Comparator): Group 3 will receive the Self Help e-Book as a comparative condition (families provided a kindle version copy of "Helping Your Anxious Child: A Step-by-Step Guide" ; Rapee, Wignall, Spence, Lyneham, & Cobham, 2008).
  Interventions: Behavioral: Self-Help E-Book
- 4: Waitlist Control (No Intervention): Group 4 will not receive any intervention, but will be randomized into an active study arm at 6 weeks.

INTERVENTIONS:
Behavioral: Anchors Away — Modular Cognitive Behavioral Therapy delivered through a mobile app.
  Arms: 1: Anchors Away
Behavioral: Parent Enhanced Anchors Away — Modular Cognitive Behavioral Therapy delivered through a mobile app. Extra modules will focus specifically on parenting skills relevant to having an anxious child.
  Arms: 2: Parent Enhanced Anchors Away
Behavioral: Self-Help E-Book — Parents will read "Helping Your Anxious Child: A Step-by-Step Guide" (Rapee, Wignall, Spence, Lyneham, & Cobham, 2008)
  Arms: 3: Self-Help E-Book

SUMMARY:
Anxiety disorders are among the most common psychological disorders, with prevalent onset in childhood and adolescence. While cognitive behavioral therapy (CBT) is considered the first-line treatment for pediatric anxiety, significant barriers remain in accessing CBT and other evidence-based treatments (EBTs), and credible self-help resources based in EBT concepts. This study evaluates a family-guided CBT game application (Anchors App), targeted to children ages 6-11 and their families, which focuses on delivering adaptive CBT-based coping skills to those who have sub-clinical to mild anxiety and related symptoms in a convenient and portable platform. Anchors App will be evaluated in two forms (standard and "parent-enhanced") in comparison to use of a self-help book or waitlist control. The rapid advancements in technology allows richer interactive capacity, content scalability, customizability, and subscription to a broader range of content, which this app capitalizes on in order to increase access to CBT skill concepts directly to pediatric stakeholder populations. If found to be effective, Anchors App has the opportunity to promote engagement of EBT concepts in every-day use through smartphone technology, and will change the landscape of mental health prevention and early intervention for children and families.

ELIGIBILITY:
Inclusion Criteria:

* Availability of mobile technology (e.g., smart phone, tablet)
* Internet access
* English language spoken in the home

Exclusion Criteria:

* Child in current or recent (last 2 months) psychotherapy
* Child currently taking psychotropic medication
* Parent or child endorsing symptom greater than 2 standard deviations above the mean on clinical measures
* Parents express feeling unable to assist child with current degree of symptoms

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Spence Children's Anxiety Scale - Parent/Child Report (SCAS) | Entry into study, 6 weeks, 12 weeks
  Parent and child report of anxiety with 6 DSM-IV criteria sub scales. Measuring change in reported anxiety levels in these 6 different domains over time.

SECONDARY OUTCOMES:
DASS-21 | Entry into study, 6 weeks, 12 weeks
  A screener for overall psychological distress of parent with sub scales assessing anxiety, depression, and stress.
Centre for Epidemiological Studies- Depression Scale for Children (CES-DC) | Entry into study, 6 weeks, 12 weeks
  A 20-item screener for childhood depression and psychological distress
Anxiety Sensitivity Index- 3 (ASI-3) | Entry into study, 6 weeks, 12 weeks
  A measure of parent anxiety sensitivity (fear of arousal-related sensations) in physical, social, and cognitive domains
Child Anxiety Sensitivity Index (CASI) | Entry into study, 6 weeks, 12 weeks
  A measure of sensitivity to symptoms of anxiety, similar to the ASI, measuring physical, social, and mental incapacitation concerns in children.
Behavioral Inhibition Instrument (BII) | Entry into study, 6 weeks, 12 weeks
  A parent-report measure of child behavioral inhibition, which has been determined to be a risk factor for later psychopathology, particularly anxiety.
Treatment Status and Parent Confidence | Entry into study, 3 weeks, 6 weeks, 12 weeks
  Self-report measure to ensure the child is not receiving outside interventions (as would disqualify them from study) and to gauge parents' confidence in managing child's symptoms
Opinion on Intervention | 6 weeks
  Self-report measure to gauge families' thoughts on user-friendliness, perceived effectiveness of intervention, and likelihood to use again or recommend to others

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn D Kriegshauser, PhD, Principal Investigator — Kansas City Center for Anxiety Treatment, P.A.; Lisa R Hale, PhD, Principal Investigator — Kansas City Center for Anxiety Treatment, P.A.; Margo Adams Larsen, PhD, Principal Investigator — Virtually Better, Inc.
Locations (1):
- Kansas City Center for Anxiety Treatment, P.A., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No